CLINICAL TRIAL: NCT00815217
Title: The Role of Lipoaspirate Injection in the Treatment of Diabetic Lower Extremity Wounds and Venous Stasis Ulcers
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: due to PI work schedule and no personnel resources
Sponsor: Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 01194
Record Dates: First submitted 2008-12-24; First posted 2008-12-29 (Estimated); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Diabetic Wounds; Venous Stasis Wounds
Keywords: Lipoaspirate; Diabetes Mellitus; Mesenchymal Stem cells; Fat grafts; venous stasis
MeSH Terms: conditions — Diabetes Mellitus; Varicose Ulcer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 lipoaspirate (Experimental): wounds which have received the lipoaspirate
  Interventions: Procedure: injection of lipoaspirate
- 2 control (Placebo Comparator): For the control wound, only the sterile injectable tumescence solution (1 liter of LR, 30 cc of 1% lidocaine, 1 ampule of 1:1,000,000 epinepherine) will be used. The solution will be injected in a similar fashion with single tunnels radially around the control wound spaced at 5-10 mm apart and approximately 3 - 5 cm in length.
  Interventions: Other: control

INTERVENTIONS:
Procedure: injection of lipoaspirate — Small volume lipoaspiration will be performed. This technique involves harvesting small amounts of fat by making a small incision in the donor site (usually the abdomen) and infiltrating 25-75cc of tumescence solution (1 liter of LR, 30 cc of 1% lidocaine, 1 ampule of 1:1,000,000 epinepherine) into the adipose layer with a blunt infiltrator. The Coleman aspiration Cannulae, approximately 2-3 mm in diameter and 15 cm in length attached with a Luer-Lok suction syringe will be used to harvest up to 100 cc of fat. Gently pulling back on the syringe provides a small amount of negative pressure to allow for aspiration into the syringe.For the intervention wound, the adipose tissue will be implanted using the infiltration Cannulae (blunt end, 7 cm- COL-17) or the both approx. 1mm in diameter. The implantation will be in single tunnels radially around each wound spaced at 5-10 mm apart and approximately 3 - 5 cm in length.
  Arms: 1 lipoaspirate
Other: control — For the control wound, only the sterile injectable tumescence solution (1 liter of LR, 30 cc of 1% lidocaine, 1 ampule of 1:1,000,000 epinepherine) will be used. The solution will be injected in a similar fashion with single tunnels radially around the control wound spaced at 5-10 mm apart and approximately 3 - 5 cm in length.
  Arms: 2 control

SUMMARY:
A prospective, single blinded randomized clinical study will be performed to determine if the injection of lipoaspirate into diabetic or venous stasis wounds promotes wound healing or wound closure at a faster rate than conventional treatment.

DETAILED DESCRIPTION:
Diabetic lower extremity wounds and venous stasis wounds are two of the most challenging, costly medical problems of our population. Moreover, the Veterans Affairs population has a very high percentage of diabetes and venous stasis wounds.

Foot ulcers are the most common reason for a diabetic patient to be admitted to the hospital, and occur in approx 25% of patients (CDC) with an average stay of 3 weeks and a cost of 25,000$/ per treatment (21,22, 23). The pathophysiology of diabetic wound healing is characterized by microcirculatory ischemia and an abnormal wound healing cascade due to glycosylated cells and proteins.

Venous stasis disease affects 10-35% of the US population (24) and is characteristically difficult to treat, recurrent and costly. The dermal microcirculation is aberrant with cellular stasis, capillary leak, edema and prone to chronic wounds. As venous pressures increase in these patients, there is microcirculatory ischemia which predisposes to wound formation.

In the skin, the normal wound healing cellular cascade mechanism acts to restore epithelial components and ends in collagen deposition and scar formation. Imperative to this process is angiogenesis, cellular signaling, and cellular mitosis. These wound healing processes can be promoted by stem cell transplantation.

It is now known that lipoaspirate obtained by standard small volume liposunction techniques contains autologous mesenchymal stem cells. We propose that autologous stem cell transplantation via lipoaspirate injection to these recalcitrant wounds could be a safe and effective treatment modality. Because the cellular derangement of both diabetic wounds and venous stasis wounds is derived from abnormal cell signaling, micro-ischemia and abnormal capillaries, stem cell treatment which can aid in angiogenesis and cellular signaling may be a treatment option which is aimed directly at the root cause of the disease.

Aim 1: A prospective, single blinded randomized clinical study will be performed to determine if the injection of lipoaspirate into diabetic or venous stasis wounds promotes wound healing or wound closure at a faster rate than conventional treatment.

Rationale: Despite considerable effort, successful healing of diabetic lower extremity wounds and venous stasis wounds remain as a difficult therapeutic challenge. We will examine whether autologous lipoaspirate injection is a safe and effective treatment option for diabetic lower extremity wounds and venous stasis wounds.

Hypothesis: Injection of lipoaspirate subcutaneously around diabetic wounds and venous stasis wounds will promote wound healing more effectively than conventional treatments.

ELIGIBILITY:
INCLUSION CRITERIA:

* Patients with diabetic lower extremity wounds or venous stasis wounds present for more than 6 months whose wounds have failed to heal with conventional medical therapy will be included.
* Only fully consentable and compliant patients who are already scheduled to undergo surgical wound treatment or wound debridement in the operating room or in clinic will be included.
* Only patients with palpable distal pulses will be included.

EXCLUSION CRITERIA:

* Patients with the following criteria will be excluded:

  * HIV + patients
  * patients on anticoagulants which cannot be stopped or corrected
  * patients with cellulitis, infection, osteomyelitis, stage III or IV ulcers, *those patients with no safe donor site availability and dialysis dependent end stage renal disease.
* Following normal operating room protocol, anticoagulants and aspirin will be stopped prior to the procedure.
* Patients will be randomly chosen to enter the intervention arm or the control arm of the study. Even social security numbers will be chosen to undergo the treatment arm and odd social security numbers will be chosen to undergo the control arm. After randomization, the control groups and the intervention groups will be analyzed to ensure that there are no statistically significant differences in patient profiles including: albumin levels, hematocrit, smoking status, and Hgb A1C values.
* Both insulin dependent and non-insulin dependent diabetic patients will be included and Hgb A1C values will be used to ensure both groups are similar.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-02; Primary Completion 2010-02 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
wound measurements, healing of wounds, pictures of wounds | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Veterans Affairs Medical Center, Washington D.C., Washington D.C., District of Columbia, United States